CLINICAL TRIAL: NCT02761460
Title: The Study of Evaluating the Efficacy and Safety of PEG-rhG-CSF in Preventing Chemotherapy-induced Neutropenia
Brief Title: The Efficacy and Safety of PEG-rhG-CSF in Preventing Chemotherapy-induced Neutropenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: wang shusen (Other)
Responsible Party: Sponsor-Investigator, wang shusen, Chief Physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-FXY-083
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEG-rhG-CSF (Experimental): PEG-rhG-CSF 6mg is given for patients Greater than or equal to 45 kg, 3mg is given for those less than 45kg 24-48 hours after chemotherapy,
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — PEG-rhG-CSF 6mg is given for patients Greater than or equal to 45 kg, 3mg is given for those less than 45kg 24-48 hours after chemotherapy

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of PEG-rhG-CSF in preventing chemotherapy-induced neutropenia

DETAILED DESCRIPTION:
Neutrophilic granulocytopenias is one of the most common and most serious complications in chemotherapy. Research shows that about 25% ~ 40% in patients receiving standard chemotherapy can appear neutropenia with fever. It can increase the risk of infection and Chemotherapy related death, and lead to the delay of chemotherapy, and maybe Reduce the curative effect of chemotherapy. RhG-CSF has widely used to prevent neutropenia, but its half-time is short, and need daily injections to maintain the effective blood drug concentration. Patients are with poor compliance, related adverse reaction and medical costs increase. At the same time, some patients appear neutropenia thought RhG-CSF is given. Therefore, how to reduce the frequency of RhG-CSF injections and more effectively prevent neutropenia more effectively, on the premise of ensure the safety of patients to achieve better effect of chemotherapy, has always been the focus of the clinical problem.

Pegylated recombinant human granulocyte-colony stimulating factor(PEG-rhG-CSF) is a first class national new drug developed by domestic pharmaceutical companies. According to some phase Ⅱand phase Ⅲ clinical trials, PEG-rhG-CSF has a good effect. The patients need only one injection for PEG-rhG-CSF each Cycle of chemotherapy, and the effect of rising white blood cell is more smoothly, and it can avoid pain of repeated injection of PEG-rhG-CSF

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent Histologically proven breast cancer
2. Patients need to accept many cycles chemotherapy alone
3. appears III/IV neutropenia after last cycle of chemotherapy, and plan in the subsequent cycle using the same chemotherapy program.
4. KPS≥70
5. Lifetime is expected to more than 3 months
6. Before enrollment,ANC≥ANC ≥1.5×109 /L,Platelet Count (PLT) ≥80×109 /L, White Blood Cell （WBC ）≥3.0×109 /L.
7. Sign Informed Consent Form （ICF）.

Exclusion Criteria:

1. There is any difficult to control infection, or within 72 h before chemotherapy received antibiotic treatment systematically
2. Any abnormal bone marrow hyperplasia and other hematopoietic function was abnormal
3. Suffer from other malignant tumor was not cured, or patients with brain metastasis
4. Total Bilirubin （TBIL）,Alanine Transminase （ALT）,Aspartate aminotransferase(AST)>2.5×ULN
5. Cr>1.5×ULN
6. Be allergic to this product or other genetically engineered e. coli sources of biological products
7. Mental or neurological disorders
8. Women with pregnancy or lactation; The childbearing age women refused to accept contraception
9. The investigators think that the person doesn't fit into the group

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2016-05-04 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the rate of Ⅲ or Ⅳ class of neutropenia | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Wang, Doctor, Study Chair — Sun Yat-sen University
Locations (1):
- Shusen Wang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided